CLINICAL TRIAL: NCT00534495
Title: Randomized Placebo Phase Study of Rilonacept in the Treatment of Systemic Juvenile Idiopathic Arthritis (RAPPORT)
Brief Title: Safety and Effectiveness of Rilonacept for Treating Systemic Juvenile Idiopathic Arthritis in Children and Young Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS) (NIH)
Responsible Party: Principal Investigator, Norman Ilowite, Chief, Division of Rheumatology, Children's Hospital at Montefiore, National Institute of Arthritis and Musculoskeletal and Skin Diseases (NIAMS)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: N01 AR070015; 268200700015C-2-0-0 (NIH); HHSN2682007000015C
Record Dates: First submitted 2007-09-24; First posted 2007-09-26 (Estimated); Results first posted 2015-12-11 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-11

CONDITIONS: Juvenile Idiopathic Arthritis
Keywords: Systemic Juvenile Idiopathic Arthritis; Juvenile Rheumatoid Arthritis; Systemic Juvenile Rheumatoid Arthritis
MeSH Terms: conditions — Arthritis, Juvenile; Rheumatoid Arthritis, Systemic Juvenile | interventions — rilonacept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Group 1 (Experimental): Loading dose of rilonacept (4.4mg/kg) at Week 0, followed by rilonacept 2.2 mg/kg/week for the remainder of the study
  Interventions: Biological: Rilonacept
- Group 2 (Placebo Comparator): Placebo for 4 weeks, followed by rilonacept loading dose (4.4mg/kg), followed by rilonacept 2.2 mg/kg/week for the remainder of the study
  Interventions: Biological: Rilonacept

INTERVENTIONS:
Biological: Rilonacept — 2.2 mg/kg subcutaneously
  Other Names: IL-1 Trap; Arcalyst

SUMMARY:
Systemic juvenile idiopathic arthritis (SJIA) is a type of arthritis that typically occurs before 16 years of age. SJIA usually involves heat, pain, swelling, and stiffness in the body's joints. It can also involve fever, rash, anemia, and inflammation in various parts of the body. Rilonacept is a drug that can reduce inflammation. The purpose of this study is to determine whether a rilonacept drug regimen initiated early is more effective than a similar rilonacept drug regimen initiated 4 weeks later when treating children and young adults with SJIA.

DETAILED DESCRIPTION:
The current standard treatment for SJIA includes nonsteroidal anti-inflammatory drugs (NSAIDS) and corticosteroids. However, in most people, NSAIDS do not completely control the disease. Also, no studies have been done to prove which medication or combination of medications is best to treat children and adolescents with SJIA. Interleukin-1 (IL-1), a protein secreted by certain cells in the body, assists in regulating immune and inflammatory responses. Too much IL-1 can be harmful and has been shown to play a role in the inflammation associated with a variety of diseases, including SJIA. Rilonacept is a drug that inhibits IL-1 activity. The purpose of this study is to determine whether a rilonacept drug regimen initiated early is more effective than a similar rilonacept drug regimen initiated 4 weeks later when treating children and young adults with SJIA. This study will also evaluate the safety of rilonacept, and various tissue samples will be collected from participants for future genetic studies.

This study will last 6 months. Participants will be randomly assigned to one of two groups:

* Group 1 participants will receive rilonacept injections at a dose of 4.4mg/kg at study entry (loading dose), then 2.2 mg/kg weekly until Week 4. At Week 4, they will receive a loading dose of placebo, followed by weekly rilonacept injections at 2.2 mg/kg for the duration of the study.
* Group 2 participants will receive placebo at study entry and then during the first 4 weeks of treatment. At Week 4, they will receive a loading dose of rilonacept injections of 4.4 mg/kg, followed by weekly rilonacept injections at a dose of 2.2 mg/kg for the duration of the study.

Participants will continue any previous corticosteroid therapy, but in tapering doses. All participants will attend study visits at Weeks 0, 2, 4, 6, 8, 10, 12, 14 and 24. Study visits will include a physical exam, joint exam, blood collection, interview, and questionnaires. Urine collection may occur for some female participants. Other evaluations may be performed by the participant's regular doctor. Throughout the study, participants will maintain at-home diaries to record fever, morning stiffness and pain, when rilonacept or placebo was taken, any side effects experienced from treatment, and any additional medications that were taken.

ELIGIBILITY:
Inclusion Criteria:

* Fulfills International League Against Rheumatism (ILAR) criteria for SJIA
* Duration of SJIA lasting at least 6 weeks since onset
* Active disease as defined by at least two joints with active disease
* Not currently receiving methotrexate OR if taking methotrexate, the dose has remained stable or has been discontinued for 4 weeks prior to screening
* Has never received certain biologics OR if previously received biologics, discontinued etanercept for at least 4 weeks prior to screening and discontinued infliximab or adalimumab for at least 8 weeks prior to screening
* Not currently receiving corticosteroids OR if taking oral corticosteroids, the dose has remained stable between 2 and 60 mg/day for at least 2 weeks prior to screening

Exclusion Criteria:

* Past treatment with anakinra, rilonacept, or other biologic IL-1 inhibitor
* Treatment with other disease-modifying antirheumatic drugs (DMARDs) including, but not limited to, azathioprine, sulfasalazine, cyclosporine, and thalidomide within 4 weeks of screening
* Treatment with leflunomide without cholestyramine washout at the end of therapy
* Treatment with cyclophosphamide within 3 months of study entry
* Treatment with tacrolimus or tocilizumab within 4 weeks of study entry
* Treatment with rituximab within 6 months of study entry
* Treatment with intravenous immunoglobulin (IVIG) within 4 weeks of screening
* Kidney disease
* AST or ALT levels more than two times the upper limit of normal
* Bilirubin levels higher than 1.5 mg/dl
* Thrombocytopenia, leukopenia, or neutropenia
* Abnormal prothrombin time (PT) and partial thromboplastin time (PTT) tests
* Low levels of plasma fibrinogen
* Evidence of chronic recurrent infection or other significant, non-SJIA illness that might interfere with study participation
* Psychological or cognitive difficulties that might interfere with study participation
* Current drug or alcohol abuse
* Anticipated poor compliance to assigned study regimen
* Participation in another clinical trial within 30 days of study entry
* Major surgical procedure within 3 months of study entry

Ages: 18 Months to 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 71 (Actual)
Dates: Start 2008-11; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Norman T. Ilowite, MD, Principal Investigator — Montefiore Medical Center
Locations (1):
- Montefiore Medical Center, The Bronx, New York, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 71 participants enrolled. 1 participant was erroneously randomized and was not included in the analysis. This patient was not exposed to study drug
Groups:
- Rilonacept: Loading dose of rilonacept (4.4mg/kg) at Week 0, followed by rilonacept 2.2 mg/kg/week followed by a placebo loading dose and then rilonacept in the long term extension phase Rilonacept: 2.2 mg/kg subcutaneously
- Placebo: Placebo loading dose followed by maintenance dose for 4 weeks, followed by rilonacept loading dose (4.4mg/kg), followed by rilonacept 2.2 mg/kg/week for the long term extension
  Rilonacept: 2.2 mg/kg subcutaneously
- Long Term Extension All Participants: All participants who benefited from rilonacept were eligible to enroll this phase and receive rilonacept 2.2mg/kg weekly
Period: Double Blind Placebo Phase Week 0-4
Arm/Group | Rilonacept | Placebo | Long Term Extension All Participants
Started | 36 | 35 | 0
Completed | 36 | 34 | 0
Not Completed | 0 | 1 | 0
Not completed — randomized in error | 0 | 1 | 0
Period: All Active Treatment Phase Week 4-24
Arm/Group | Rilonacept | Placebo | Long Term Extension All Participants
Started | 36 | 34 | 0
Completed | 32 | 25 | 0
Not Completed | 4 | 9 | 0
Not completed — Adverse Event | 1 | 0 | 0
Not completed — Lack of Efficacy | 1 | 7 | 0
Not completed — Lost to Follow-up | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 1 | 0
Period: Long Term Ext. Phase Week 24-month 21
Arm/Group | Rilonacept | Placebo | Long Term Extension All Participants
Started | 0 | 0 | 40
Completed | 0 | 0 | 29
Not Completed | 0 | 0 | 11
Not completed — Adverse Event | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 5
Not completed — Withdrawal by Subject | 0 | 0 | 3
Not completed — non compliance | 0 | 0 | 2

BASELINE CHARACTERISTICS:
Groups:
- Rilonacept: Loading dose of rilonacept (4.4mg/kg) at Week 0, followed by rilonacept 2.2 mg/kg/week for the remainder of the study
  Rilonacept: 2.2 mg/kg subcutaneously
- Placebo: Placebo for 4 weeks, followed by rilonacept loading dose (4.4mg/kg), followed by rilonacept 2.2 mg/kg/week for the remainder of the study
  Rilonacept: 2.2 mg/kg subcutaneously
- Total: Total of all reporting groups
Arm/Group | Rilonacept | Placebo | Total
Number analyzed (Participants) | 36 | 35 | 71
Age, Continuous [Mean (Standard Deviation); unit: years] | 9.5 (4.6) | 10.5 (4.4) | 10 (4.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 23 | 46
  Male | 13 | 12 | 25
Race/Ethnicity, Customized [Number; unit: Participants] — Black ,white and Other are races Hispanic and Non-Hispanic are ethnicities. All patients were counted twice.
  Participants
    Black | 5 | 7 | 12
    White | 25 | 23 | 48
    Other | 6 | 5 | 11
    Hispanic | 7 | 5 | 12
    Non-Hispanic | 29 | 30 | 59
Disease Duration [Mean (Standard Deviation); unit: years] | 2.6 (3.6) | 2.6 (3.1) | 2.6 (3.4)
No.of joints with active disease [Mean (Standard Deviation); unit: joints] | 11.7 (9.6) | 10.5 (7.6) | 11.1 (8.6)
Prior medications [Number; unit: participants]
  Corticosteroids | 30 | 33 | 63
  Methotrexate | 21 | 26 | 47
  Leflunomide | 1 | 2 | 3
  Infliximab | 5 | 6 | 11
  Etanercept | 12 | 16 | 28
  Abatacept | 5 | 4 | 9
  Anakinra | 13 | 13 | 26
  unknown Anakinra | 4 | 4 | 8
Disease characteristics in the past [Number; unit: participants]
  Incomplete Macrophage Activation Syndrome | 1 | 3 | 4
  Complete Macrophage Activation Syndrome | 1 | 1 | 2
  Serositis | 9 | 8 | 17
  Systemic JIA rash | 32 | 33 | 65

OUTCOME MEASURES:

1. Primary Outcome: Time to Response to Treatment, as Determined by a Modified JIA ACR30 Requiring no Fever, Coupled With a Requirement for Corticosteroid Taper in Participants Who Are Taking Corticosteroids
Time Frame: At Week 12
Measure: Median (Inter-Quartile Range); unit: weeks
Arm/Group | Rilonacept | Placebo
Number analyzed (Participants) | 36 | 35
weeks | 4 [2 to 10] | 8 [6 to NA] — not estimable too few events

2. Secondary Outcome: Number of Participants With Response as Determined by JIA ACR50 and JIA ACR70
Time Frame: At Week 4 and week 12
Population: Participants in the study at week 4 (rilonacept 35 and placebo 33).Participants in the study at week 12 ( Rilonacept 33 and placebo 29).
Measure: Number; unit: participants
Arm/Group | Rilonacept | Placebo
Number analyzed (Participants) | 35 | 33
participants
  week 4 ,ACR 50 | 21 | 10
  week 12, ACR 50 | 26 | 13
  week 4 ,ACR 70 | 21 | 10
  week 12,ACR 70 | 28 | 19

3. Secondary Outcome: Pediatric Quality of Life Inventory
Description: Visual Analog Score (0-100 mm) 0 very well , 100 very poor
Time Frame: At Weeks 4, 12 and 24
Population: At Week 4 ,36 Rilonacept and 34 Placebo patient. At week 12, Rilonacept 33 patients and Placebo 29.At baseline Rilonacept 36 and Placebo 35 participants.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Rilonacept | Placebo | Week 24- All Subjects
Number analyzed (Participants) | 36 | 35 | 57
units on a scale
  week 4 | 12 [3 to 23] | 34 [15 to 67] | NA [NA to NA] — At week 24 both arms were combined
  week 12 | 3.5 [0 to 17] | 8 [2 to 38] | NA [NA to NA] — At week 24 both arms were combined
  week 24 | NA [NA to NA] — At week 24 both arms were combined | NA [NA to NA] — At week 24 both arms were combined | 7 [1 to 29]
  baseline | 49.5 [33 to 65] | 53.0 [28 to 68] | NA [NA to NA] — At week 24 both arms were combined

4. Secondary Outcome: Physical Function as Determined by Childhood Health Assessment Questionnaire ( CHAQ)
Description: Childhood Health Assesment Questionairre dissability index (C-HAQ)-DI, Disability Index Calculation:
  The index is calculated by adding the scores for each of the categories and dividing by the number of categories answered. This gives a score in the 0 to 3.0 range. lower is better
Time Frame: At Weeks 12 and 24
Population: 36 Rilonacept and 35 placebo at baseline , 36 Rilonacept and 34 placebo at week 4, 33 Rilonacept and 29 placebo at week 12, and 57 combined at week 24.
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | Rilonacept | Placebo | Week 24- All Subjects
Number analyzed (Participants) | 36 | 35 | 57
units on a scale
  week 4 | 0.43 [0.00 to 1.13] | 0.88 [0.38 to 1.63] | NA [NA to NA] — Groups were combined at week 24
  week 12 | 0.25 [0.00 to 0.88] | 0.25 [0.00 to 1.25] | NA [NA to NA] — Groups were combined at week 24
  week 24 | NA [NA to NA] — Groups were combined at week 24 | NA [NA to NA] — Groups were combined at week 24 | 0.13 [0.00 to 1.00]
  baseline | 1.00 [0.75 to 1.63] | 1.25 [0.50 to 1.63] | NA [NA to NA] — Groups were combined at week 24

5. Secondary Outcome: Number of Participants With Presence of Systemic Features ( Fever, Rash)
Time Frame: At Weeks 4, 12 and 24
Population: At week 4 ,Rilonacept 36 and Placebo 34 participants , at week 12 , Rilonacept 33 and 29 Placebo participants , and at week 24 combined group with 57 participants, at baseline Rilonacept 36 and Placebo 35 participants.
Measure: Number; unit: participants
Arm/Group | Rilonacept | Placebo | Week 24- All Subjects
Number analyzed (Participants) | 36 | 35 | 57
participants
  Fever at week 4 | 3 | 5 | NA — data not collected
  Rash at week 4 | 3 | 8 | NA — data not collected
  Fever at week12 | 4 | 1 | NA — data not collected
  Rash at week 12 | 3 | 1 | NA — data not collected
  week 24 Fever | NA — not collected | NA — not collected | NA — not collected
  week 24 Rash | NA — both groups were combined at 24 weeks | NA — both groups were combined at 24 weeks | 4
  baseline Fever | 10 | 6 | NA — data not collected
  beseline Rash | 15 | 15 | NA — data not collected

6. Primary Outcome: Number of Serious Adverse Events,Adverse Events, Infections, Development of MAS
Time Frame: At Weeks 0- 24
Measure: Number; unit: events
Arm/Group | Rilonacept | Placebo | Long Term Extension 24 Weeks to 21 Months
Number analyzed (Participants) | 36 | 35 | 40
events
  Serious Adverse Events | 4 | 2 | 8
  Adverse Events | 98 | 186 | 110
  Infections | 27 | 31 | 37
  MAS | 1 | 0 | 0

ADVERSE EVENTS:
Groups:
- Rilonacept Week (0-4); Rilonacept Week (4-24): Loading dose of rilonacept (4.4mg/kg) at Week 0, followed by rilonacept 2.2 mg/kg/week for the remainder of the study
  Rilonacept: 2.2 mg/kg subcutaneously
- Placebo Week (0-4); Placebo Week (4-24): Placebo for 4 weeks, followed by rilonacept loading dose (4.4mg/kg), followed by rilonacept 2.2 mg/kg/week for the remainder of the study
  Rilonacept: 2.2 mg/kg subcutaneously
Arm/Group | Rilonacept Week (0-4) | Placebo Week (0-4) | Rilonacept Week (4-24) | Placebo Week (4-24) | Long Term Extension 24 Weeks to 21 Months
Serious Adverse Events (participants affected / at risk) | 1/36 | 1/35 | 3/35 | 1/33 | 6/40
Other Adverse Events (participants affected / at risk) | 9/36 | 19/35 | 27/35 | 28/33 | 28/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Rilonacept Week (0-4) (N=36) | Placebo Week (0-4) (N=35) | Rilonacept Week (4-24) (N=35) | Placebo Week (4-24) (N=33) | Long Term Extension 24 Weeks to 21 Months (N=40)
Juvenile Arthritis (Musculoskeletal and connective tissue disorders) | 1 | 1 | 0 | 1 | 1
Abnormal Liver Function Test (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Pyrexia (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Variccela (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Viral uper respiratory tract infestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Mental status Changes (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Pericarditis (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Pharingitis,Streptoccocal (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Gastroenteritis ,Salmonela (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Histiocytosis,hematophagic (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Rilonacept Week (0-4) (N=36) | Placebo Week (0-4) (N=35) | Rilonacept Week (4-24) (N=35) | Placebo Week (4-24) (N=33) | Long Term Extension 24 Weeks to 21 Months (N=40)
Abdominal pain ,upper (Gastrointestinal disorders) | 1 | 2 | 3 | 1 | 0 — Adverse events
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 2 | 6 | 1 — Adverse events
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 2 | 3 | 2 — Adverse events
Headache (General disorders) | 1 | 6 | 1 | 4 | 3 — Adverse events
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 2 | 3 — Adverse events
Pharyngitis,Streptococcal (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2 | 4 — Adverse events
Pyrexia (Infections and infestations) | 0 | 1 | 5 | 1 | 1 — Adverse events
Rash (Immune system disorders) | 2 | 1 | 1 | 3 | 1 — Adverse events
Upper Respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 5 | 9 | 2 — Adverse events
Vomiting (Gastrointestinal disorders) | 1 | 2 | 1 | 2 | 4 — Adverse events
injection site reaction (General disorders) | 2 | 7 | 2 | 3 | 0
Body temperature increased (Investigations) | 0 | 2 | 3 | 2 | 0
Urinary tract infections (Infections and infestations) | 0 | 0 | 3 | 1 | 0
Fatigue (General disorders) | 0 | 1 | 1 | 2 | 0
Non Cardiac chest pain (General disorders) | 0 | 3 | 1 | 4 | 0
Pain (General disorders) | 0 | 1 | 0 | 2 | 2
Rhinorea (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 2 | 4 | 0
Nasal Congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 2 | 0
dyspnea (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 3 | 1 | 3
diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 2 | 0
Joint swelling (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 2 | 3
dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 2 | 0
Erythema (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 2 | 0
Dizziness (Nervous system disorders) | 0 | 1 | 0 | 2 | 0
Blood fibrinogen dicreased (Investigations) | 0 | 0 | 0 | 4 | 0
Alanine amino transferase Increased (Investigations) | 0 | 0 | 0 | 0 | 2
Aspartate Amino transferase increased (Investigations) | 0 | 0 | 0 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No